CLINICAL TRIAL: NCT01310075
Title: Bioprosthetic Mesh to Expand the Lower Pole in Tissue Expander Reconstruction: A Blinded, Prospective, Randomized, Controlled Trial
Brief Title: Bioprosthetic Mesh to Expand the Lower Pole in Tissue Expander Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-0324; NCI-2011-01477 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: Mastectomy; Bioprosthetic Mesh; Breast Reconstruction; Tissue Expander; Alloderm; Surgimend
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alloderm Mesh (Experimental): Alloderm Mesh - 6 x 12 cm piece or 6 x 16 cm piece is trimmed into a semicircle and sewn into the inframammary fold using vicryl. The smooth side is placed against the implant.
  Interventions: Device: Alloderm
- Surgimend Mesh (Experimental): Surgimend Mesh - 10 x 15 cm piece of fenestrated material is sewn to the fold, curved side along the fold, using vicryl suture.
  Interventions: Device: Surgimend
- Control (no mesh) (No Intervention)

INTERVENTIONS:
Device: Alloderm — 6 x 12 cm piece or 6 x 16 cm piece is trimmed into a semicircle and sewn into the inframammary fold using vicryl. The smooth side is placed against the implant.
  Arms: Alloderm Mesh
Device: Surgimend — 10 x 15 cm piece of fenestrated material is sewn to the fold, curved side along the fold, using vicryl suture.
  Arms: Surgimend Mesh

SUMMARY:
The goal of this clinical research study is to learn if the complication rate and post-surgical appearance differ based on what type of mesh is used for breast reconstruction surgery.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be randomly assigned (as in the roll of a dice) to receive Surgimend mesh or Alloderm mesh.

Breast Reconstruction Surgery:

All techniques of the breast reconstruction surgery are considered to be standard of care. You will be given a separate consent form to sign that explains the procedure and risks in more detail.

Data Collection:

Information about you will be collected, including your age, height, weight, breast size, past medical and smoking history, tumor size and location, and the surgical method used for the breast reconstruction surgery.

Information about the breast reconstruction surgery, such as what type of expanders are used, the surgical methods, and your recovery from the surgery will also be collected.

Follow-Up Visits:

About 1 week after the breast reconstruction surgery is complete, you will come in for a follow-up visit and the surgical team will check the surgery incision site and tissue used for the breast reconstruction surgery for any possible complications.

About 2 weeks after the breast reconstruction surgery, the expansion process will begin, as long as you do not have any complications that would prevent beginning the expansion process. During the expansion process, the surgeon will adjust the tissue expanders to stretch the area under the skin and muscle to make room for a breast implant(s).

After you begin the expansion process, you will return to the clinic 1 time each week for additional expansion until the desired size is reached. During each of the expansion process visits, you will be checked for any side effects, including fluid build up and infection.

After the expansion process is complete, you will return to the clinic 3 months later to receive your implant(s). About 1 to 12 months after you receive the implant(s), you will return to the clinic and 5 photographs will be taken to evaluate the appearance of the new implant(s). The photographs will be taken of the front, right and left sides of the implant(s) site and will be taken against a blue background. Your private areas will be covered (as much as possible). Your confidentiality will be protected at all times. You will not be identifiable personally from the discussion or presentation of the data. Unique study numbers will be assigned to the photographs.

Length of Study:

Your participation on this study will be over after you have received your permanent breast implant(s) and the photographs have been taken.

This is an investigational study.

Up to 398 patients will take part in this study. All will be enrolled at the MD Anderson main campus or one of the MD Anderson regional care centers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing immediate tissue expander reconstruction following mastectomy by any of the surgeon co-investigators are eligible for the study.
2. Patients 18 years of age or older are eligible for the study.
3. Patients undergoing skin-sparing mastectomy utilizing bioprosthetic mesh are eligible for the study.
4. Patients who have not undergone autologous tissue breast reconstruction and intend to undergo implant only breast reconstruction.
5. Patients who intend to remain under the MDACC surgeon's care until completion of the reconstruction.

Exclusion Criteria:

1. Patients with prior radiation to the breast/chest wall of the ipsilateral breast .
2. Patients who cannot be effectively reconstructed without the use of bioprosthetic mesh.
3. Patients who are current smokers.
4. Patients requiring additional intra-operative skin resections of greater than 1cm beyond the skin edge as a result of mastectomy flap devascularization.
5. Patients who have a history of breast tissue expander or implant placement.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Clemens, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study began enrollment on 04/15/2011 and was closed to enrollment on 12/08/2015. All recruitment done at the University of Texas MD Anderson Cancer Center.
Groups:
- Arm 1- Surgimend: Surgimend Mesh - 10 x 15 cm piece of fenestrated material is sewn to the fold, curved side along the fold, using vicryl suture.
- Arm 2-Alloderm: Alloderm Mesh - 6 x 12 cm piece or 6 x 16 cm piece is trimmed into a semicircle and sewn into the inframammary fold using vicryl. The smooth side is placed against the implant.
  Device: Alloderm 6 x 12 cm piece or 6 x 16 cm piece is trimmed into a semicircle and sewn into the inframammary fold using vicryl. The smooth side is placed against the
Period: Overall Study
Arm/Group | Arm 1- Surgimend | Arm 2-Alloderm
Started | 45 | 45
Completed | 31 | 35
Not Completed | 14 | 10
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 10 | 7
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Surgimend
- Arm 2: Alloderm
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 31 | 35 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 31 | 61
  >=65 years | 1 | 4 | 5
Age, Continuous [Mean (Full Range); unit: years] | 48.06 [30 to 70] | 48.69 [31 to 71] | 48.39 [30 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 35 | 66
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 24 | 29 | 53
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 26 | 29 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 35 | 65
  Guatemala | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complications After Tissue Expander Replacement With Implant
Time Frame: through study completion, an average of 1 year
Population: Of the 90 randomized participants, 66 (74%) were evaluable for the primary measure
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 31 | 35
participants | 10 | 10

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/35
Serious Adverse Events (participants affected / at risk) | 3/31 | 2/35
Other Adverse Events (participants affected / at risk) | 8/31 | 18/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=31) | Arm 2 (N=35)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Delayed wound healing (Skin and subcutaneous tissue disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=31) | Arm 2 (N=35)
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 3 | 8
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 2
Hematoma (Vascular disorders) | 0 | 1
Seroma (Vascular disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Delayed wound healing (Skin and subcutaneous tissue disorders) | 2 | 0
Wound dehiscensence (Skin and subcutaneous tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT01310075/Prot_SAP_000.pdf